CLINICAL TRIAL: NCT04604184
Title: BI 764198 Efficacy and Safety in Prevention/Progression of ARDS and ARDS-related Complications Secondary to COVID-19 (ACTION ON COVID-19)
Brief Title: ACTION ON COVID-19: A Study to Test Whether BI 764198 Helps Lung Health of People Hospitalised With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1434-0009; 2020-003211-96 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-10-27 (Actual); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 764198 treatment group (Experimental)
  Interventions: Drug: BI 764198
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 764198 — BI 764198
  Arms: BI 764198 treatment group
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults with COVID-19 infection who are in hospital and receive oxygen. Participants need to be 50 years of age or older and need to be at risk of further worsening of their condition.

The purpose of the study is to find out whether a medicine called BI 764198 helps people with COVID-19 infection and breathing problems. BI 764198 may prevent cell death and swelling of the lung tissue and therefore help patients with COVID-19 infection.

Participants are put into 2 groups by chance. One group of participants gets BI 764198 capsules and the other group gets placebo capsules. The placebo capsules look exactly like the BI 764198 capsules but do not contain any medicine. Participants take 1 capsule per day.

Participants are in the study for about a month. At study end, doctors compare the 2 groups for the number of patients that are alive and do not need mechanical breathing support. During the study, the doctors collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* SARS-CoV-2 infection positive confirmed by PCR or approved point-of-care test
* A score of 5 (hospitalised; oxygen by mask or nasal prongs) or 6 (hospitalised; oxygen by non-invasive ventilation or high flow), but not previously ≥7, on the WHO Clinical Progression Scale.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must abstain from male female sex or must use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly during hospitalisation for at least 7 days after last trial drug intake

Exclusion Criteria:

* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >5 × the upper limit of normal (ULN).
* Known active infection with HIV or hepatitis B or C.
* Pulmonary oedema/respiratory failure due to cardiogenic insult.
* Previous to hospitalisation, on long-term oxygen therapy.
* A confirmed baseline prolongation of QTc interval to greater than 450 ms in males or 470 ms in females according to the Bazett formula, or any other relevant ECG finding at screening, or concomitant use of medication prolonging QT interval.
* Stage 4 severe chronic kidney disease or requiring dialysis (i.e., eGFR <30 mL/min/1.73 m2).

History of the following cardiac conditions:

* Myocardial infarction within 3 months prior to the first dose
* Unstable angina
* History of clinically significant long QT features on electrocardiogram (ECG) or history of familial long QT

  * Anticipated transfer/discharge to another hospital or care facility other than their place of residence
  * Further exclusion criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (7):
  - University of California Irvine, Orange, California
  - Rapides Regional Medical Center, Alexandria, Louisiana
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Providence Regional Medical Center, Everett, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
- Brazil (5):
  - Hospital Luxemburgo, Belo Horizonte
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Hospital Ernesto Dornelles, Porto Alegre
  - Hospital Regional Hans Dieter Schmidt, Santa Catarina
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
- Chile (2):
  - Hospital Padre Alberto Hurtado, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- Mexico (3):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Hospital General de Culiacán "Dr. Bernardo J. Gastellum", Culiacán
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Puerto Rico (2):
  - Hospital Auxilio Mutuo, Hato Rey
  - Hospital Municipal de San Juan, Rio Piedras
- Spain (6):
  - Hospital A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Espases, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Ware LB, Soleymanlou N, McAuley DF, Estrada V, Diaz GA, Lacamera P, Kaste R, Choi W, Gupta A, Welte T. TRPC6 inhibitor (BI 764198) to reduce risk and severity of ARDS due to COVID-19: a phase II randomised controlled trial. Thorax. 2023 Aug;78(8):816-824. doi: 10.1136/thorax-2022-219668. Epub 2023 Apr 6. PMID 37024277
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomised, placebo-controlled, double-blind, proof-of-concept exploratory trial was to evaluate the efficacy and safety of BI 764198, an inhibitor of the transient receptor potential subtype C6 (TRPC6), compared to placebo in reducing risk or severity of acute respiratory distress syndrome (ARDS) in patients hospitalised for coronavirus disease appeared in 2019 (COVID-19).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 764198 Treatment Group: Subjects who were hospitalised for infection with SARS-CoV-2, the virus that causes COVID-19 received BI 764198, oral or, only if needed, per nasogastric intubation once per day starting on Day 1, with a treatment duration of up to 28 days.
- Placebo: Subjects who were hospitalised for infection with SARS-CoV-2, the virus that causes COVID-19 received Placebo, oral or, only if needed, per nasogastric intubation once per day starting on Day 1, with a treatment duration of up to 28 days.
Period: Overall Study
Arm/Group | BI 764198 Treatment Group | Placebo
Started | 67 | 66
Treated | 65 | 64
Completed | 47 | 47
Not Completed | 20 | 19
Not completed — Adverse Event | 5 | 5
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Not treated | 2 | 2
Not completed — Due to sponsor decision | 9 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Transfer to healthcare | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS included all patients (pts) in randomized set (RS) who received at least 1 dose of trial drug, comprised 129 pts (85.4%). Of all pts randomised, number (%) of pts not treated was similar in BI 764198 (2/67 pts [3.0%]) and placebo group (2/66 pts [3.0%]). The 4 pts excluded from FAS discontinued trial before receiving treatment for following reasons: pt's withdrawal (n=2), meeting an exclusion criterion (n=1), and clinical worsening (n=1).
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 764198 Treatment Group | Placebo | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (8.3) | 63.6 (7.9) | 63.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 41 | 39 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 35 | 74
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 12
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 3 | 3 | 6
  White | 53 | 47 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Free of Mechanical Ventilation
Description: Percentage of patients alive and free of mechanical ventilation at Day 29 is presented.
  One patient had no creatinine at baseline value and was therefore excluded from the statistical analysis (N=128).
Time Frame: At Day 29
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Percentage of patients | 83.1 | 87.5
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Test type: Other; p = 0.3232, Regression, Logistic; includes treatment, age, severity grade and creatinine at baseline, duration of symptoms before hospitalisation as covariates; Risk Difference (RD) = -5.39, 95% CI 2-sided [-16.08 to 5.30]

2. Secondary Outcome: Percentage of Patients Alive and Discharged Free of Oxygen Use
Description: Percentage of patients alive and discharged free of oxygen use is presented. One patient had no creatinine at baseline value and was therefore excluded from the statistical analysis (N=128).
Time Frame: At Day 29
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Percentage of patients | 75.4 | 82.8
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Test type: Other; p = 0.1274, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -9.86, 95% CI 2-sided [-22.54 to 2.82]

3. Secondary Outcome: Percentage of Patients With Occurrence of Any Component of Composite: In-hospital Mortality or Intensive Care Unit (ICU) Admission or Mechanical Ventilation
Description: Percentage of patients with occurrence of any component of composite: In-hospital mortality or intensive care unit (ICU) admission or mechanical ventilation is presented.
  Efficacy endpoint meets when a patient has occurrence of any component of composite: In-hospital mortality or intensive care unit (ICU) admission or mechanical ventilation at Day 29.
  One patient had no creatinine at baseline value and was therefore excluded from the statistical analysis (N=128).
Time Frame: At Day 29
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Percentage of patients | 26.2 | 23.4
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Test type: Other; p = 0.6828, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 2.66, 95% CI 2-sided [-10.11 to 15.43]

4. Secondary Outcome: Time to Clinical Improvement of at Least 2 Points (From Randomisation) on the World Health Organization Clinical Progression Scale, Discharge From the Hospital, or Considered Fit for Discharge
Description: Meets when improvement of at least 2 points on World Health Organization (WHO) Clinical Progression Scale (CPS), discharge from hospital, fit for discharge (score 0, 1, 2, 3 on CPS), whichever comes first.
  WHO CPS: 0. Uninfected; no viral RNA detected; 1. Asymptomatic; viral RNA detected; 2. Symptomatic; independent; 3. Symptomatic; assistance needed; 4. Hospitalised; no oxygen therapy; 5. Hospitalised; oxygen by mask or nasal prongs; 6. Hospitalised; oxygen by non-invasive ventilation or high flow; 7. Intubation + mechanical ventilation, partial pressure of oxygen/fraction of inspired oxygen (pO2/FiO2) ≥150 or oxygen saturation/FiO2 (SpO2/FiO2) ≥200; 8. Mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors; 9. Mechanical ventilation pO2/FiO2 <150 + vasopressors, dialysis, extracorporeal membrane oxygenation (ECMO); 10. Death Only patients with event were analysed. One patient had no creatinine at baseline value, therefore excluded from statistical analysis (N=128).
Time Frame: Up to Day 29
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Days | 9 [6 to 24] | 7 [5 to 10]
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Test type: Other; p = 0.0445, Regression, Cox; Covariates are treatment, age, severity grade and creatinine at baseline and duration of symptoms before hospitalization; Rate Ratio = 0.67, 95% CI 2-sided [0.46 to 0.99]

5. Secondary Outcome: Number of Ventilator Free Days
Description: Number of ventilator free days by Day 29 is presented. One patient had no creatinine at baseline value and was therefore excluded from the statistical analysis (N=128).
Time Frame: Up to Day 29
Population: Full Analysis Set (FAS): FAS included all patients (pts) in randomized set (RS) who received at least 1 dose of trial drug, comprised 129 pts. Only pts with non-missing results were included. Of all pts randomised, number of pts not treated was similar in BI 764198 (2/67 pts) and placebo group (2/66 pts). The 4 pts excluded from FAS discontinued trial before receiving treatment for following reasons: pt's withdrawal (n=2), meeting an exclusion criterion (n=1), and clinical worsening (n=1).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Days | 24.12 (8.81) | 25.08 (7.85)
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Test type: Other; p = 0.5526, ANCOVA; Fixed effects of treatment, age, severity grade and creatinine at baseline and duration of symptoms before hospitalisation as covariates; Mean Difference (Net) = -0.80, 95% CI 2-sided [-3.47 to 1.87], Standard Error of Mean 1.35 — Difference = covariate adjusted BI 764198 - covariate adjusted Placebo

6. Secondary Outcome: Percentage of Mortality at Day 15, 29, 60 and 90
Description: Percentage of mortality is presented. One patient had no creatinine at baseline value and was therefore excluded from the statistical analysis (N=128).
Time Frame: At Day 15, 29, 60 and 90
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | BI 764198 Treatment Group | Placebo
Number analyzed (Participants) | 65 | 64
Percentage of patients
  Day 15 | 6.2 | 1.6
  Day 29 | 12.3 | 7.8
  Day 60 | 15.4 | 7.8
  Day 90 | 16.9 | 7.8
Statistical Analysis 1: Comparison: BI 764198 Treatment Group vs Placebo; Day 15; Test type: Other; p = 0.0995, Regression, Logistic; Includes treatment, age, severity grade and creatinine at baseline, and duration of symptoms before hospitalisation as covariates; Risk Difference (RD) = 5.32, 95% CI 2-sided [-1.01 to 11.65]
Statistical Analysis 2: Comparison: BI 764198 Treatment Group vs Placebo; Day 29; Test type: Other; p = 0.1992, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Risk Difference (RD) = 6.06, 95% CI 2-sided [-3.19 to 15.31]
Statistical Analysis 3: Comparison: BI 764198 Treatment Group vs Placebo; Day 60; Test type: Other; p = 0.0709, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Risk Difference (RD) = 8.93, 95% CI 2-sided [-0.76 to 18.62]
Statistical Analysis 4: Comparison: BI 764198 Treatment Group vs Placebo; Day 90; Test type: Other; p = 0.0412, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Risk Difference (RD) = 10.35, 95% CI 2-sided [0.41 to 20.28]

ADVERSE EVENTS:
Time Frame: From first administration of the study drug to end of study, 90 days in total.
Description: Full Analysis Set (FAS): FAS included all patients (pts) in randomized set (RS) who received at least 1 dose of trial drug, comprised 129 pts (85.4%). Of all pts randomised, number (%) of pts not treated was similar in BI 764198 (2/67 pts [3.0%]) and placebo group (2/66 pts [3.0%]). The 4 pts excluded from FAS discontinued trial before receiving treatment for following reasons: pt's withdrawal (n=2), meeting an exclusion criterion (n=1), and clinical worsening (n=1).
Arm/Group | BI 764198 Treatment Group | Placebo
All-Cause Mortality (participants affected / at risk) | 11/65 | 5/64
Serious Adverse Events (participants affected / at risk) | 19/65 | 17/64
Other Adverse Events (participants affected / at risk) | 10/65 | 12/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 764198 Treatment Group (N=65) | Placebo (N=64)
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 4 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Deep vein thrombosis (Vascular disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Right ventricular dilatation (Cardiac disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Citrobacter infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Distributive shock (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 764198 Treatment Group (N=65) | Placebo (N=64)
Constipation (Gastrointestinal disorders) | 4 | 6
Electrocardiogram QT prolonged (Investigations) | 3 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypotension (Vascular disorders) | 4 | 5
Tachycardia (Cardiac disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
This trial was terminated early following the recommendation of a Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04604184/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04604184/SAP_001.pdf